CLINICAL TRIAL: NCT02025192
Title: A Phase 1b, Open-label Study to Assess the Safety and Tolerability of Tucatinib (ONT-380) Combined With Capecitabine and Trastuzumab, Alone and in Combination in HER2+ Metastatic Breast Cancer
Brief Title: A Study of Tucatinib (ONT-380) Combined With Capecitabine and/or Trastuzumab in Patients With HER2+ Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONT-380-005
Record Dates: First submitted 2013-12-17; First posted 2013-12-31 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: HER2 Positive Metastatic Breast Cancers
Keywords: ONT-380; Capecitabine; Trastuzumab; Xeloda; Herceptin; HER2 positive breast cancer; Breast cancer; ARRY-380; Tucatinib
MeSH Terms: conditions — Breast Neoplasms | interventions — tucatinib; Capecitabine; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tucatinib (ONT-380) in combination with capecitabine (Experimental)
  Interventions: Drug: Tucatinib; Drug: Capecitabine
- Tucatinib (ONT-380) in combination with trastuzumab (Experimental)
  Interventions: Drug: Tucatinib; Drug: Trastuzumab
- Tucatinib (ONT-380) combined with capecitabine and trastuzumab (Experimental)
  Interventions: Drug: Tucatinib; Drug: Capecitabine; Drug: Trastuzumab

INTERVENTIONS:
Drug: Tucatinib — Administered twice per day, orally.
  Other Names: ONT-380
Drug: Capecitabine — 1000mg/m^2 administered twice per day, orally in Days 1-14 of each 21-day cycle.
  Other Names: Xeloda
  Arms: Tucatinib (ONT-380) combined with capecitabine and trastuzumab; Tucatinib (ONT-380) in combination with capecitabine
Drug: Trastuzumab — Administered at a loading dose of 8 mg/kg IV followed by 6 mg/kg once every 21 days.
  Other Names: Herceptin
  Arms: Tucatinib (ONT-380) combined with capecitabine and trastuzumab; Tucatinib (ONT-380) in combination with trastuzumab

SUMMARY:
The purpose of this study is to determine the maximal tolerated dose (MTD) or recommended phase 2 dose (RP2D) of tucatinib (ONT-380) and to assess the safety and tolerability of tucatinib (ONT-380) combined with capecitabine alone, trastuzumab alone and with both capecitabine and trastuzumab in patients with HER2+ metastatic breast cancer.

DETAILED DESCRIPTION:
This is a study of tucatinib (ONT-380) given in combination with capecitabine alone, trastuzumab alone and with both capecitabine and trastuzumab in patients with HER2+ metastatic breast cancer.

This study will use a 3+3 dose escalation design to evaluate escalating dose levels of tucatinib (ONT-380) in each of these three combinations in order to identify the maximal tolerated dose/recommended phase 2 dose (MTD/RP2D) of tucatinib (ONT-380). The MTD/RP2D of tucatinib (ONT-380) to be used in combination with either capecitabine alone (Combination 1) or trastuzumab alone (Combination 2) will be determined prior to evaluating tucatinib (ONT-380) in combination with both capecitabine and trastuzumab (Combination 3). If Combination 1 and Combination 2 are found to be tolerable, then tucatinib (ONT-380) will be evaluated in Combination 3, using the lowest MTD/RP2D or other SMC-recommended dose of tucatinib (ONT-380) determined for either of the two drug combinations. This will be followed by enrollment of an expansion cohort of patients treated at the MTD/RP2D for Combination 3. Additional expansion cohorts for either Combination 1 (tucatinib (ONT-380) and capecitabine) or Combination 2 (tucatinib (ONT-380) and trastuzumab) may also be enrolled.

Capecitabine will be given twice per day orally at 1000 mg/m^2 on Days 1-14 of each 21-day cycle. Trastuzumab will be given as a loading dose of 8 mg/kg IV followed by 6 mg/kg once every 21 days. However, a loading dose of trastuzumab will not be given to patients who have received trastuzumab within 4 weeks of the first study dose of trastuzumab. These patients will receive trastuzumab at 6 mg/kg each cycle, including Cycle 1. Trastuzumab may also be given on a weekly basis at 2 mg/kg IV q 7 days, but only in the circumstance that trastuzumab infusion has been delayed, and weekly infusions are required to resynchronize the cycle length to 21 days, after discussion with the medical monitor. Trastuzumab infusion rates will be per institutional guidelines. Tucatinib (ONT-380) will be given twice per day orally at a dose dependent upon the dosing cohorts to which the patient is enrolled.

There will be 3-6 evaluable patients enrolled in each cohort in the dose escalation phase, unless that dose is found to be intolerable prior to completion of enrollment. At least 6 evaluable patients are to be treated at a dose level in order for an MTD/RP2D to be determined.

Provided that only seven dose cohorts are needed for dose escalation and only the expansion cohort for Combination 3 is enrolled, up to 66 evaluable patients may be enrolled. Additional patients may be enrolled if additional expansion cohorts are opened.

ELIGIBILITY:
Inclusion Criteria

* Metastatic breast cancer, documented as HER2+ by fluorescence in situ hybridization (FISH) and/or 3+ staining by immunohistochemistry (IHC).
* Progressive disease, with a history of prior treatment with both trastuzumab and T-DM1 (unless deemed intolerant to or ineligible for T-DM1 by the investigator) for metastatic disease.
* If female and of child-bearing potential, has negative pregnancy test within 14 days prior to treatment.
* If a sexually active male or a sexually active female of child-bearing potential, agrees to use dual (two concurrent) forms of medically accepted contraception from the time of consent until 6 months after the last dose of ONT-380, capecitabine, or trastuzumab, whichever is longest.
* Must have target or non-target lesions as per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
* All toxicity related to prior cancer therapies must have resolved to ≤ Grade 1, with the following exceptions: alopecia; neuropathy, which must have resolved to ≤ Grade 2; and congestive heart failure (CHF), which must have been ≤ Grade 1 in severity at the time of occurrence and must have resolved completely.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at screening.
* In the opinion of the Investigator, life expectancy > 6 months.
* Adequate hematologic function as defined by:

  1. Hemoglobin ≥ 9 g/dL
  2. Absolute neutrophil count (ANC) ≥ 1000 cells/μL
  3. Platelets ≥ 100,000/μL
* Adequate hepatic function as defined by the following:

  1. Total bilirubin ≤ 1.5 X upper limit of normal (ULN), unless a known history of Gilbert's disease
  2. Transaminases (aspartate aminotransferase/serum glutamic oxaloacetic transaminase [AST/SGOT] and alanine aminotransferase/serum glutamic pyruvic transaminase [ALT/SGPT]) ≤ 2.5 X ULN (< 5 X ULN if liver metastases are present)
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 X ULN unless on medication known to alter INR and aPTT.
* Creatinine clearance ≥ 50 mL/min.
* Left ventricular ejection fraction (LVEF) must be within institutional limits of normal as assessed by echocardiogram (ECHO) or multiple-gated acquisition scan (MUGA) documented within 4 weeks prior to first dose of study drug.

Exclusion Criteria

* Medical, social, or psychosocial factors that, in the opinion of the Investigator, could impact safety or compliance with study procedures.
* Patient is breastfeeding.
* Previous treatment with any experimental agent within 14 days or five half-lives of study treatment, whichever is greater.
* Previous treatment with trastuzumab or other antibody-based therapy within three weeks of starting study treatment or with chemotherapy or hormonal cancer therapy within two weeks of starting study treatment.
* Previous treatment with cumulative dose of doxorubicin > 360 mg/m2 or previous treatment with another anthracycline with cumulative dose equivalent to > 360 mg/m2 doxorubicin.
* Previous treatment with:

  1. Capecitabine for metastatic disease at any time, for patients assigned to cohorts using capecitabine plus ONT-380 (Combination 1) or capecitabine plus trastuzumab plus ONT-380 (Combination 3). However, patients who have previous treatment with capecitabine for metastatic disease are eligible for enrollment into cohorts using trastuzumab plus ONT-380 (Combination 2). Patients who have received capecitabine for adjuvant or neoadjuvant treatment at least 12 months prior to starting study treatment are eligible to enroll into all cohorts (Combination 1, 2, or 3).
  2. Any small molecule HER2 inhibitors including (but not limited to) lapatinib, neratinib, or afatinib within the last 4 weeks prior to initiation of study therapy.
* CNS disease:

  1. Patients with leptomeningeal disease are excluded.
  2. Dose escalation and expansion cohorts: Patients with symptomatic CNS metastases are excluded. Patients with treated CNS metastases or untreated asymptomatic CNS metastases not requiring immediate local therapy may be eligible. Enrollment of patients with metastases must be approved by the study medical monitor.
  3. Optional CNS disease expansion cohorts: Patients with untreated asymptomatic CNS metastases not requiring immediate local therapy or patients with progressive CNS disease following local therapy may be eligible with medical monitor approval.
* History of allergic reactions to compounds of similar chemical or biological composition to capecitabine (for patients assigned to Combination 1 or 3 only), trastuzumab (for patients assigned to Combination 2 or 3 only), or ONT-380, except for a history of Grade 1 or Grade 2 Infusion Related Reaction to trastuzumab, which has been successfully managed.
* Patients with uncorrectable electrolyte abnormalities.
* Known to be HIV positive. HIV testing is not required for those patients who are not known to be positive.
* Known carrier of Hepatitis B and / or Hepatitis C (whether active disease or not).
* Known liver disease, autoimmune hepatitis, or sclerosing cholangitis.
* Inability to swallow pills or any significant gastrointestinal diseases, which would preclude adequate absorption of oral medications.
* Use of a strong CYP3A4 inhibitor or inducer within three elimination half-lives of the inhibitor or inducer prior to the start of study treatment.
* Use of a strong CYP2C8 inducer or inhibitor within three elimination half-lives of the inducer or inhibitor prior to the start of study treatment. (See Appendix F).
* Radiotherapy within 14 days of first dose of ONT-380; patient must have recovered from acute effects of radiotherapy to baseline.
* Known impaired cardiac function or clinically significant cardiac disease such as ventricular arrhythmia requiring therapy, congestive heart failure, and uncontrolled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg on antihypertensive medications).
* Myocardial infarction or unstable angina within 6 months prior to the first dose of study drug.
* Patient with known dihydropyrimidine dehydrogenase deficiency (for patients assigned to Combination 1 or 3 only).
* Patient requiring warfarin therapy with known history of difficulty in management of maintaining INR within therapeutic range. Patients on warfarin may be included if on a stable dose with a therapeutic INR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-12-31 (Actual); Primary Completion 2017-10-03 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to approximately 4 years
Severity of adverse events | Up to approximately 4 years

SECONDARY OUTCOMES:
Incidence of clinical lab abnormalities (hematology, chemistry, liver function tests, coagulation, urinalysis) | Up to approximately 4 years
Severity of clinical lab abnormalities (hematology, chemistry, liver function tests, coagulation, urinalysis) | Up to approximately 4 years
Frequency of dose reductions in tucatinib (ONT-380 | Up to approximately 4 years
Frequency of dose reductions in capecitabine | Up to approximately 4 years
Plasma concentrations of tucatinib (ONT-380) and metabolite | 26 months
Plasma concentrations of capecitabine and metabolites | 26 months
Objective response rate (ORR) | 26 months
  Objective response (OR) will be defined as a best response of complete response (CR) or partial response (PR). The ORR will be calculated as the proportion of patients in the Efficacy Evaluable Patient Set who achieve an objective response.
Duration of response | 26 months
Disease control rate | 26 months
  Disease control will be defined as a best response of CR, PR, or stable disease (SD). The DCR will be calculated as the proportion of patients in the Efficacy Evaluable Patient Set who achieve disease control.
Clinical benefit rate (CBR) | 26 months
  Clinical benefit will be defined as a best response of CR, PR, or SD for ≥ 6 months. The CBR will be calculated as the proportion of patients in the Efficacy Evaluable Patient Set who achieve clinical benefit.
Progression-free survival (PFS) | Up to 6 years
  PFS will be defined as the time from first dose of study drug until documentation of disease progression or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: JoAl Mayor, PharmD, BCOP, Study Director — Seagen Inc.; Corinna Palanca-Wessels, MD, PhD, Study Director — Seagen Inc.
Locations (5):
- United States (5):
  - University of Colorado, Aurora, Colorado
  - Providence Cancer Center, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Northwest Medical Specialties, Tacoma, Washington

REFERENCES:
- [Derived] Zhang D, Taylor A, Zhao JJ, Endres CJ, Topletz-Erickson A. Population Pharmacokinetic Analysis of Tucatinib in Healthy Participants and Patients with Breast Cancer or Colorectal Cancer. Clin Pharmacokinet. 2024 Oct;63(10):1477-1487. doi: 10.1007/s40262-024-01412-0. Epub 2024 Oct 5. PMID 39368039
- [Derived] Murthy R, Borges VF, Conlin A, Chaves J, Chamberlain M, Gray T, Vo A, Hamilton E. Tucatinib with capecitabine and trastuzumab in advanced HER2-positive metastatic breast cancer with and without brain metastases: a non-randomised, open-label, phase 1b study. Lancet Oncol. 2018 Jul;19(7):880-888. doi: 10.1016/S1470-2045(18)30256-0. Epub 2018 May 24. PMID 29804905